CLINICAL TRIAL: NCT06047184
Title: A Phase I, Open, Multicenter Study of BEBT-209 in Women With Advanced Breast Cancer
Brief Title: Phase I Study of BEBT-209 in Women With Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BeBetter Med Inc (Industry)
Collaborators: Hunan Cancer Hospital (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-209-P01
Record Dates: First submitted 2023-09-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Advanced Breast Cancer
Keywords: BEBT-209; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — Letrozole; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Dose escalation phase: 6 dose levels are carried out, the starting dose of BEBT-209 is set to 25mg/day, and the accelerated titration method combined with the "3+3" mode is used for climbing research.
  Phase Ib: According to the pharmacokinetics, safety and preliminary efficacy of BEBT-209 in the dose escalation phase, one dose was selected for the BEBT-209 monotherapy group, two doses were selected for the combination with letrozole group, and two doses were selected for the combination with fulvestrant group, and all five groups were continuously administered until disease progression or unacceptable toxicity or patient withdrawal or death.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Monotherapy group 1 (Experimental): BEBT-209 capsules, 25mg once daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules
- Monotherapy group 2 (Experimental): BEBT-209 capsules, 25mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules
- Monotherapy group 3 (Experimental): BEBT-209 capsules, 50mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules
- Monotherapy group 4 (Experimental): BEBT-209 capsules, 75mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules
- Monotherapy group 5 (Experimental): BEBT-209 capsules, 100mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules
- Monotherapy group 6 (Experimental): BEBT-209 capsules, 150mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules
- BEBT-209 combined with the letrozole group 1 (Experimental): BEBT-209 capsules, 100mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Letrozole tablets, 2.5mg each time, once a day for 4 weeks, 4 weeks as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules; Drug: Letrozole tablets
- BEBT-209 combined with the letrozole group 2 (Experimental): BEBT-209 capsules, 75mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Letrozole tablets, 2.5mg each time, once a day for 4 weeks, 4 weeks as a treatment cycle.
  Interventions: Drug: BEBT-209 capsules; Drug: Letrozole tablets
- BEBT-209 combined with the Fulvestrant Group 1 (Experimental): BEBT-209 capsules, 75mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Fulvestrant, injection, 500mg each time, 1 time on day 1 and day 15 of the first cycle, and once on the first day of each cycle from the second cycle, 4 weeks as a treatment cycle
  Interventions: Drug: BEBT-209 capsules; Drug: Fulvestrant
- BEBT-209 combined with the Fulvestrant Group 2 (Experimental): BEBT-209 capsules, 100mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Fulvestrant, injection, 500mg each time, 1 time on day 1 and day 15 of the first cycle, and once on the first day of each cycle from the second cycle, 4 weeks as a treatment cycle
  Interventions: Drug: BEBT-209 capsules; Drug: Fulvestrant

INTERVENTIONS:
Drug: BEBT-209 capsules — BEBT-209 capsules, 25mg once daily, or 25mg, 50mg, 75mg, 100mg, 150mg each time, twice daily, were administered continuously for 3 weeks and discontinued for 1 week, and 4 weeks were used as a treatment cycle.
  Other Names: KCBT-0191
Drug: Letrozole tablets — Letrozole tablets, 2.5mg each time, once a day for 4 weeks, 4 weeks as a treatment cycle.
  Other Names: Femara
  Arms: BEBT-209 combined with the letrozole group 1; BEBT-209 combined with the letrozole group 2
Drug: Fulvestrant — Fulvestrant, injection, 500mg each time, 1 time on day 1 and day 15 of the first cycle, and once on the first day of each cycle from the second cycle, 4 weeks as a treatment cycle
  Other Names: FASLODEX
  Arms: BEBT-209 combined with the Fulvestrant Group 1; BEBT-209 combined with the Fulvestrant Group 2

SUMMARY:
This clinical study includes a dose escalation trial of BEBT-209 monotherapy in HR +/HER2- advanced breast cancer patients and a Phase 1b trial of BEBT-209 as a single therapy, in combination with letrozole, and in combination with fulvestrant in ER +/HER2- advanced breast cancer in women. To evaluate the safety, tolerability, pharmacokinetic profile, and preliminary efficacy of BEBT-209 as a single therapy, in combination with letrozole, and in combination with fulvestrant. To determine the recommended dose for late clinical studies of monotherapy or combination therapy in patients with HR +/HER2- advanced breast cancer.

DETAILED DESCRIPTION:
* Dose escalation phase: To conduct approximately 6 dose levels, with a starting dose of 25 mg/day of BEBT-209, and subsequent dose groups were first dose escalated at 100%, with dose escalation at 50% for subsequent dose groups if one drug-related Grade 2 nonhematologic or Grade 3 hematologic toxicity was identified and dose-limiting toxicity was not reached. If one dose limiting toxicity was identified and the maximum tolerated dose was not reached, dose escalation was performed at 33% for the subsequent dose groups.
* Phase Ib of BEBT-209 as single therapy, in Combination with Letrozole, in Combination with Fulvestrant: According to the pharmacokinetics, safety and preliminary efficacy of BEBT-209 in the dose escalation phase, one dose was selected for the BEBT-209 monotherapy group, two doses were selected for the combination with letrozole group, and two doses were selected for the combination with fulvestrant group, and all five groups were continuously administered until disease progression or unacceptable toxicity or patient withdrawal or death. Late phase clinical trials were conducted as appropriate based on preliminary safety tolerability, pharmacokinetics, and preliminary efficacy results from Phase 1b.

Participants will need to understand the requirements and risks of the trial, sign an informed consent form, accept the dosing regimen required by the trial protocol, and follow the investigator's guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old;
2. Confirmed HR +/HER2- breast cancer in women with evidence of focal recurrence or metastasis not amenable to curative surgical resection or radiation therapy.
3. Menstrual status:

   3.1 Subjects enrolled in the dose escalation phase, Phase Ib combined with letrozole, combined with fulvestrant first-line therapy were required to be female patients who achieved menopausal status or were treated with LHRH agonists; 3.2 Subjects enrolled in Phase Ib monotherapy and combined fulvestrant second-line/third-line therapy are required to be postmenopausal, premenopausal/ perimenopausal, and amenorrheic women;

   Menopausal status(note 2) is defined as having met any of the following:
   * Prior bilateral oophorectomy;
   * Age≥ 60 years old
   * Age < 60 years, Spontaneous amenorrhea ≥ 12 months and blood follicle-stimulating hormone (FSH) and estradiol (E2) levels within the postmenopausal range (in conjunction with reference ranges at each site) in the absence of chemotherapy, tamoxifen, toremifene, or ovarian castration within the past year;
   * Patients < 60 years of age who were taking tamoxifen or toremifene had blood follicle-stimulating hormone (FSH) and estradiol (E2) levels within the postmenopausal range on two consecutive occasions (in conjunction with reference ranges at each site);
   * Not meeting the above criteria for menopause is considered premenopausal or perimenopausal; Note 2:Premenopausal/perimenopausal female patients agree to use concomitant luteinizing hormone-releasing hormone (LHRH agonist) and start treatment with LHRH agonist at least 28 ± 2 days before the start of the first dose of study drug can be considered to meet inclusion criteria 3.1 (if LHRH agonist has been used for ≥ 21 days but < 26 days before the first dose, hormone levels are eligible can be considered to meet inclusion criteria 3.1) ;
4. Prior Therapy( Note 3):

   4.1 Patients who have failed standard therapy or for whom standard therapy is not applicable are required for the dose escalation phase; 4.2 Phase IB monotherapy group: patients who have previously failed antiestrogen therapy and received at least 1 chemotherapy regimen; 4.3 The stage IB combined letrozole group required no previous first-line treatment for focal recurrent or metastatic ER + breast cancer; 4.4 Prior therapy in the Stage IB combined fulvestrant arm must have met one of the following: 4.4.1 Premenopausal/perimenopausal/postmenopausal patients can be enrolled, and premenopausal/perimenopausal patients are required to use luteinizing hormone-releasing hormone (LHRH agonist) at the same time; 4.4.2 Progression confirmed by imaging during or within 12 months after discontinuation of adjuvant endocrine therapy (AI or TAM); 4.4.3 Progression confirmed by imaging during or within one month after discontinuation of endocrine therapy for the first recurrence and metastasis; 4.4.4 Patients in the relapse or metastatic stage are allowed to receive no more than one line of chemotherapy in addition to endocrine therapy.

   Note 3: The number of lines of therapy and corresponding menstrual status definitions refer to the Ribociclib Phase 3 Clinical Study (NCT02422615), the abemaciclib Phase 2 Clinical Study (Clin Cancer Res. 2017 September 01; 23 (17): 5218 - 5224), and the Palbociclib in Combination with Fulvestrant Clinical Study (NCT02738866).
5. Measurable lesions as defined by RECIST V.1.1 or osteolytic bone metastases only as judged by the investigator based on clinical presentation. Tumor lesions previously treated with radiotherapy or other local therapy were considered measurable only if disease progression at the treatment site was clearly documented after completion of treatment.
6. ECOG score of 0-2.
7. Have adequate organ and bone marrow function, defined as follows: ANC≥1,500/mm^3（1.5 x 10^9 /L）； Platelet ≥ 100,000/mm^3 (100 x10

   ^9 /L）； hemoglobin≥ 9 g/dL (90 g/L); Both ALT or AST ≤ 2.5×ULN, and ALT or AST ≤ 5.0×ULN in liver metastasis; Total bilirubin (TBIL) ≤ 1.5×ULN, 3.0×≤ULN in liver metastasis; Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 60 mL/min (according to the Cockcroft and Gault formula).
8. Resolution of all acute toxicities from prior anticancer therapy or surgical procedures to baseline severity or NCICTCAE version 5.0 ≤ Grade 1 (except alopecia or other toxicities that, in the opinion of the investigator, pose no safety risk to the patient).
9. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to starting study drug and be willing to use a medically recognized highly effective form of birth control (eg, intrauterine device, contraceptive pill, or condom) during the study and for 1 month after the last dose of study drug.
10. Willing to sign the informed consent form after thorough understanding.

Exclusion Criteria:

1. combined with any other malignancy (except adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ).
2. symptomatic, advanced patients who have disseminated to the viscera and are at risk of life-threatening complications in the short term (patients with visceral crisis); inflammatory breast cancer.
3. Known or symptomatic active CNS metastases characterized by clinical symptoms, cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, and/or progressive growth.
4. Major surgery, chemotherapy, radiation therapy, any investigational agent, or other anticancer therapy within 4 weeks prior to the first dose.
5. Patients who have received the following treatments within 7 days prior to study entry: drugs known to be potent inhibitors/inducers of CYP3A4; drugs known to significantly prolong the QT interval.
6. previous treatment with CDK4/6 inhibitors.
7. Patients previously treated with fulvestrant and everolimus cannot be enrolled in cohorts 4 and 5.
8. QTc interval > 480 msec (based on the average of three screening electrocardiograms [ECGs]); a history or confirmed family history of long QT syndrome; a history of clinically significant ventricular arrhythmias, or current use of antiarrhythmic drugs or a defibrillator device implanted to treat ventricular arrhythmias.
9. Uncontrolled electrolyte disturbances that may affect the effects of QTc prolonging drugs.
10. previous myocardial infarction, severe/unstable angina pectoris, NCICTCAE version 5.0 grade ≥ 2 sustained arrhythmia, atrial fibrillation of any grade, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism);
11. active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or any upper gastrointestinal surgery including gastrectomy; known malabsorption syndrome or other conditions that may impair absorption of BEBT-209.
12. Known history of hypersensitivity or suspected symptoms of hypersensitivity to any component of letrozole, fulvestrant, BEBT-209 capsules.
13. Clinically significant active infections including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS) -related diseases. Active hepatitis B was defined as having positive hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg) and HBV DNA ≥ 2000 IU/ml (equivalent to 104 copies/ml); active hepatitis C was defined as having HCV RNA above the lower limit of detection.
14. Other serious acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk of study participation or increase the risk associated with study drug administration, or interfere with study results, as well as other conditions that, in the opinion of the investigator, would make the patient inappropriate for participation in this study.
15. Recent active suicidal ideation or behavior.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
MTD | 4 weeks
  Maximum tolerated dose
DLT | 4 weeks
  Dose-limiting toxicity

SECONDARY OUTCOMES:
ORR | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Objective response rate
CBR | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  clinical benefit rate
PFS | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  progression-free survival
DOR | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Duration of response
Cmax | Day 1 and Day 21 of cycle 1 before and within 48 hours after administration (each cycle is 28 days)
  Peak Plasma Concentration
Tmax | Day 1 and Day 21 of cycle 1 before and within 48 hours after administration (each cycle is 28 days)
  Time of peak Plasma Concentration
t1/2 | Day 1 and Day 21 of cycle 1 before and within 48 hours after administration (each cycle is 28 days)
  Half-life of plasma drug concentrations
AUC0-48h | Day 1 and Day 21 of cycle 1 before and within 48 hours after administration (each cycle is 28 days)
  Area under the blood concentration time curve from 0 to 48 hours after administration
AUC0-last | Day 1 and Day 21 of cycle 1 before and within 48 hours after administration (each cycle is 28 days)
  Area under the blood concentration time curve from time zero to the last dose
CL/F | Day 1 and Day 21 of cycle 1 before and within 48 hours after administration (each cycle is 28 days)
  Apparent total plasma clearance
Vd | Day 1 and Day 21 of cycle 1 before and within 48 hours after administration (each cycle is 28 days)
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Quchang Ouyang, Phd, Principal Investigator — Hunan Cancer Hospital; Shouman Wang, Phd, Principal Investigator — Xiangya Hospital of Central South University
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan